CLINICAL TRIAL: NCT01190033
Title: STUDY OF THE EFFICACY OF NEUROLYSIS IN FUNCTIONAL RECOVERY FROM CHRONIC NONSPECIFIC LOW BACK PAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Alexandre F. Cristante, PhD., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIZT2010; iot 803 (Other: institutional research committee)
Record Dates: First submitted 2010-08-05; First posted 2010-08-27 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neurolysis (Active Comparator): In this intervention the neurotome will be connected
  Interventions: Procedure: neurolysis
- Neurotome OFF (Placebo Comparator): neurotome not raised
  Interventions: Device: Neurotome OFF

INTERVENTIONS:
Device: Neurotome OFF — In this intervention the neurotome will be unconnected.
  Arms: Neurotome OFF
Procedure: neurolysis — In this procedure the neurotome will be connected
  Arms: Neurolysis

SUMMARY:
This is a prospective, randomized, double-blind, placebo-controlled study. In an initial phase, 100 patients with chronic low back pain will be included in this study. The patients will be recruited through magazines and newspapers to take part in a screening for treatment of low back pain. This screening will involve the evaluation of data such as history and physical examination to classify the patient in the group of nonspecific low back pain, excluding patients with neurological alterations and the so-called Red-Flags.

Procedures After the initial screening the patients will undergo diagnostic blocks of the medial branch of lumbar vertebrae L2, L3, L4 , L5 and of the first sacral vertebra (S1) with lidocaine and control with distilled water. The patients that present more than 50% of pain improvement, evaluated by the Likert scale after 30 minutes will form the study group, while the patients that do not present pain improvement with lidocaine or that present pain improvement with distilled water will be excluded.

The medial branch block consists of the insertion of a 90mm, 25-gauge needle through the skin with radioscopic control up to the medial branch topography. Infusion of 1ml of 2% lidocaine should be performed in each medial branch of the abovementioned vertebrae. Control is executed in the same manner yet with infusion of 1ml of distilled water.

Through the use of the diagnostic block we will have 40 patients selected for the second phase of the study. Once defined the study group should be evaluated before the procedure through the Oswestry, Roland Morris, SF-36 and VAS questionnaires.

In the second phase of the study the patients will be randomized. The random division into two groups will be performed through a computerized program of random numbers. The randomization result will be kept in matt sealed envelopes to guarantee secrecy of the allocation. The neurolysis procedure will be carried out in the first group, consisting of 20 patients, and the placebo or sham procedure with the second group, also with 20 patients.

The neurolysis procedure will be carried out under sterile conditions, with the patient lying prone and with the neurotome insertion sites anesthetized with 2ml of 1% lidocaine. The neurotome (Smith & Nephew - RF) will be used for the procedure. The neurotome is a radiofrequency apparatus mounted on a 10cm electrode type 22 needle with a 5mm exposure tip. The neurotome should be introduced percutaneously in a manner similar to that adopted in the medial branch block through radioscopic control. The temperature of the electrode after its placement in the correct position is then raised to 80 °C for 90 seconds. Two neurotomies should be performed for each facet, one proximally and the other distally, due to double innervation of each facet. In the patients of the placebo group the procedure will be the same only the temperature of the neurotome will not be raised. This will be performed in a blind manner, as before starting the procedure, the surgeon will show the assistant who turns the device on or not the envelope containing the patient's group (placebo or neurotomy), yet the surgeon will not be informed whether the device has been turned on or not, having to perform the procedure in the same manner in both groups.

The patients will then be reevaluated in the first month, 3 months after, 6 months after and 12 months after the procedure. The assessors will not be informed of the group to which the patient belongs, and the same scales performed in the preoperative period will be used here.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of lumbar pain in a patient with age between 20 and 60 years.
* present clinical complaints of low back pain for 3 months or more.
* present pain of moderate to severe intensity: visual analogue scale (VAS) > 4.

Exclusion Criteria:

* patients that develop a profile compatible with specific low back pain during treatment.
* patients that request their withdrawal from the study at any time.
* patients that develop an allergy to the medication used.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Pain Evaluation | The Patients will be evaluated 1 week before surgery
  Pain Scores on the Visual Analog Scale
Pain Evaluation | The Patients will be evaluated one month after surgery
  Pain Scores on the Visual Analog Scale
Pain Evaluation | The Patients will be evaluated three months after surgery
  Pain Scores on the Visual Analog Scale
Pain Evaluation | The Patients will be evaluated six months after surgery
  Pain Scores on the Visual Analog Scale
Pain Evaluation | The Patients will be evaluated one year after surgery
  Pain Scores on the Visual Analog Scale

SECONDARY OUTCOMES:
Disability evaluation | The Patients will be evaluated one week before surgery
  The Oswestry disability questionnaire has been designed to give us information as to how the back or leg pain is affecting the ability to manage in everyday life.
Medial Block Improvement | one day after the medial branch block
  likert five-level scale is a scale for evaluation of improvement:
  * 0-30% improvement - no improvement
  * 30-50% improvement - moderate improvement
  * 50-80% improvement - good improvement
  * 80-100% improvement - no pain to evaluate the improvement after the medial branch block
Health Status | The Patients will be evaluated one week before surgery
  The Roland-Morris Questionnaire (RMQ) is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale.
Disability evaluation | The Patients will be evaluated one month after surgery
  The Oswestry disability questionnaire has been designed to give us information as to how the back or leg pain is affecting the ability to manage in everyday life.
Disability evaluation | The Patients will be evaluated three month after surgery
  The Oswestry disability questionnaire has been designed to give us information as to how the back or leg pain is affecting the ability to manage in everyday life.
Disability evaluation | The Patients will be evaluated six month after surgery
  The Oswestry disability questionnaire has been designed to give us information as to how the back or leg pain is affecting the ability to manage in everyday life.
Disability evaluation | The Patients will be evaluated one year after surgery
  The Oswestry disability questionnaire has been designed to give us information as to how the back or leg pain is affecting the ability to manage in everyday life.
Health Status | The Patients will be evaluated one month after surgery
  The Roland-Morris Questionnaire (RMQ) is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale.
Health Status | The Patients will be evaluated three month after surgery
  The Roland-Morris Questionnaire (RMQ) is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale.
Health Status | The Patients will be evaluated six month after surgery
  The Roland-Morris Questionnaire (RMQ) is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale.
Health Status | The Patients will be evaluated one year after surgery
  The Roland-Morris Questionnaire (RMQ) is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Orthopedics and Traumatology of the U.S.P, São Paulo, São Paulo, Brazil